CLINICAL TRIAL: NCT00578695
Title: THE BALANCE Study: Treatment of Hyponatremia Based on Lixivaptan in NYHA Class III/IV Cardiac Patient Evaluation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CardioKine Inc. (Industry)
Collaborators: Cardiokine Biopharma, LLC (Industry); Biogen (Industry)
Responsible Party: Cardiokine, Ink, Cardiokine, Ink
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CK-LX3401
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2010-11

CONDITIONS: Hyponatremia
Keywords: Hyponatremia; Serum Sodium; Fluid Overload; Heart Failure; Acute Heart Failure; Vasopressin Antagonist
MeSH Terms: conditions — Hyponatremia; Edema; Heart Failure | interventions — lixivaptan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Experimental): Lixivaptan
  Interventions: Drug: lixivaptan
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: lixivaptan — Oral Capsule
  Arms: Active
Drug: Placebo — Oral Capsule
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety and efficacy of lixivaptan in the treatment of hyponatremia in patients with congestive heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 18 years of age or older with hyponatremia and hospitalized for congestive heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 652 (Actual)
Dates: Start 2007-01; Primary Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To determine whether lixivaptan can effectively and safely produce an increase in serum sodium from Baseline in heart failure subjects with hyponatremia and volume overload. Effects on body weight and other clinical measures will be evaluated. | 60 days

CONTACTS AND LOCATIONS:
Locations (237):
- United States (92):
  - Research Site 1, Birmingham, Alabama
  - Research Site 1, Mobile, Alabama
  - Research Site 1, Bakersfield, California
  - Research Site 1, Banning, California
  - Research Site 1, Glendale, California
  - Research Site, Glendale, California
  - Research Site 1, Los Angeles, California
  - Research Site 1, Mission Viejo, California
  - Research Site 1, Roseville, California
  - Research Site 1, San Diego, California
  - Research Site 1, Aurora, Colorado
  - Research Site 1, Newark, Delaware
  - Research Site 1, Washington D.C., District of Columbia
  - Research Site 1, Bay Pines, Florida
  - Research Site 1, Fort Lauderdale, Florida
  - Research Site 1, Gainesville, Florida
  - Research Site 1, Jacksonville, Florida
  - Research Site 1, Lakeland, Florida
  - Research Site 1, Miami, Florida
  - Research Site 1, Port Charlotte, Florida
  - Research Site 1, Tampa, Florida
  - Research Site 1, Atlanta, Georgia
  - Research Site 1, Bannockburn, Illinois
  - Research Site 1, Chicago, Illinois
  - Research Site 1, Maywood, Illinois
  - Research Site 1, Normal, Illinois
  - Research Site 1, North Chicago, Illinois
  - Research Site 1, Oak Lawn, Illinois
  - Research Site 1, Peoria, Illinois
  - Research Site 1, Munster, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Research Site 1, Iowa City, Iowa
  - Research Site 1, Louisville, Kentucky
  - Research Site 1, New Orleans, Louisiana
  - Research Site 1, Slidell, Louisiana
  - Research Site 1, Baltimore, Maryland
  - Research Site 1, Boston, Massachusetts
  - Research Site 1, Burlington, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site 1, Detroit, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - Research Site 1, Petoskey, Michigan
  - Research Site 1, Traverse City, Michigan
  - Research Site 1, Duluth, Minnesota
  - Research Site 1, St Louis, Missouri
  - Research Site 1, Lincoln, Nebraska
  - Research Site 1, Concord, New Hampshire
  - Research Site 1, Hackensack, New Jersey
  - Siant Barnabas Medical Center, Livingston, New Jersey
  - Research Site 1, Morristown, New Jersey
  - Research Site 1, Newark, New Jersey
  - Research Site 1, Orange, New Jersey
  - Research Site 1, Paramus, New Jersey
  - Research Site 1, Jamaica, New York
  - Research Site, New York, New York
  - Research Site 1, Northport, New York
  - Research Site 1, Stony Brook, New York
  - Research Site 1, The Bronx, New York
  - Research Site 1, Valhalla, New York
  - Research Site 1, Winston-Salem, North Carolina
  - Research Site 1, Cincinnati, Ohio
  - Research Site 1, Columbus, Ohio
  - Research Site 1, Fairfield, Ohio
  - Research Site, Fairfield, Ohio
  - Research Site 1, Middletown, Ohio
  - Research Site 1, Toledo, Ohio
  - Research Site 1, Oklahoma City, Oklahoma
  - Research Site 2, Oklahoma City, Oklahoma
  - Research Site 1, Tulsa, Oklahoma
  - Research Site 1, Springfield, Oregon
  - Research Site 1, Beaver, Pennsylvania
  - Research Site 1, Camp Hill, Pennsylvania
  - Research Site 1, Danville, Pennsylvania
  - Research Site 1, Pittsburgh, Pennsylvania
  - Research Site1, Sayre, Pennsylvania
  - Research Site 1, Sellersville, Pennsylvania
  - Research Site 1, Chattanooga, Tennessee
  - Research Site 1, Germantown, Tennessee
  - Research Site 1, Nashville, Tennessee
  - Research Site 1, Amarillo, Texas
  - Research Site 1, Dallas, Texas
  - Research Site 1, Galveston, Texas
  - Research Site 1, Houston, Texas
  - Research Site 1, Lubbock, Texas
  - Research Site 1, Temple, Texas
  - Research Site 1, Tyler, Texas
  - Research Site 1, Chesapeake, Virginia
  - Research Site 2, Richmond, Virginia
  - Research Site 1, Richmond, Virginia
  - Research Site 1, Seattle, Washington
  - Research Site 1, Beloit, Wisconsin
  - Research Site 1, Madison, Wisconsin
- Argentina (13):
  - Research Site, Buenos Aires, Argentina
  - Research Site 1, Buenos Aires, Argentina
  - Research Site 1, Cerrientes, Argentina
  - Research Site 1, Provincia de Buenos Aires, Argentina
  - Research Site 1, Provincia de Misiones, Argentina
  - Research Site 1, Provincia de Santa Fe, Argentina
  - Research Site 1, San Miguel de Tucumán, Argentina
  - hospital Interzonal General de Agudos, "Eva Peron" (HIGA), San Martín, Buenos Aires
  - Research Site, Ciudad Autonomo de Buenos Aires, Galvan
  - Research Site, Rosario, Santa Fe Province
  - Research Site, Buenos Aires
  - Hospital Militar Central H Gral. 601 "Cirujano Mayor Dr. Cosme Argerich", Buenos Aires
  - Hospital de Clinicas "Jose de San Martin", Buenos Aires
- Canada (11):
  - Research Site 1, Kitchener, Ontario
  - Research Site 1, Ottawa, Ontario
  - Research Site 1, Scarborough Village, Ontario
  - Research Site 1, Toronto, Ontario
  - Research Site 1, Montreal, Quebec
  - Research Site 1, Saint-Jérôme, Quebec
  - Research Site 1, Sherbrooke, Quebec
  - Research Site 1, Manitoba
  - Research Site 1, New Brunswick
  - Research Site 1, Québec
  - Research Site 1, Vancouver
- Chile (8):
  - Research Site 1, Antofagasta, Chile
  - Research Site 1, Concepción, Chile
  - Research Site 1, Orosno, Chile
  - Research Site 1, Santiago, Chile
  - Research Site, Temuco, Chile
  - Research Site 1, Viña del Mar, Chile
  - Hospital de Puerto Montt, Port Montt
  - Research Site, Santiago
- Czechia (9):
  - Research Site 1, Havlíčkův Brod
  - Research Site 1, Kladno
  - Research Site 1, Kroměříž
  - Research Site 1, Liberec
  - Research Site 1, Městec Králové
  - Research Site 1, Ostrava
  - Research Site 1, Prague
  - Research Site 1, Příbram
  - Research Site 1, Znojmo
- Germany (18):
  - Research Site 1, Bad Krozingen
  - Research Site 1, Bad Nauheim
  - Research Site 1, Bad Segeberg
  - Research Site 1, Berlin
  - Research Site 1, Bonn
  - Research Site 1, Coburg
  - Research Site 1, Dresden
  - Research Site 1, Göttingen
  - Research Site 1, Greifswald
  - Research Site 1, Hamburg
  - Research Site 1, Hanover
  - Research Site 1, Jena
  - Research Site 1, Karisbad
  - Research Site 1, Konstanz
  - Research Site 1, Leipzig
  - Research Site 1, Regensburg
  - Research Site 1, Rostock
  - Research Site 1, Soest
- India (17):
  - Research Site, Secunderabad, Andhra Pradesh
  - Research Site, Mogappair, Chennai
  - Research Site, Naranpura, Gujarat
  - Research Site, Panjagutta, Hyderabad
  - Research Site 1, Coimbatore, India
  - Research Site 1, Madhya Pradesh, India
  - Research Site 1, Maharashtra, India
  - Research Site 1, Maharastra, India
  - Research Site 1, Rajasthan, India
  - Research Site, Bangalore, Karnataka
  - Research Site, College Road, Nashik
  - Shree Saibaba Heart Institute and Research Centre, Shalimar, Nashik
  - Sir Ganga Ram Hospital, New Delhi, New Delhi
  - Research Site, Bikaner
  - Research Site, Mumbai
  - Research Site, New Delhi
  - Sri Ramachandra Medical College of research Institute, Tamul Nadu
- Israel (10):
  - Research Site 1, Beersheba, Israel
  - Research Site, Haifa, Israel
  - Research Site 1, Holon, Israel
  - Research Site, Jerusalem, Israel
  - Research Site 1, Jerusalem, Israel
  - Research Site 1, Petah Tkva, Israel
  - Research Site 1, Safed, Safed
  - Research Site 1, Tel Aviv, Tel Aviv
  - Research Site 1, Haifa
  - Research Site 1, Jerusalem
- Italy (15):
  - Research Site, Brescia, Italy
  - Research Site 1, Piacenza, Italy
  - Research Site 1, Ravenna, Italy
  - Research Site 1, Pavia, Pavia
  - Research Site 1, Torino, Torino
  - Research Site 1, Bologna
  - Research Site 1, Cecina
  - Research Site 1, Cortina
  - Research Site 1, Genova
  - Research Site 1, Milan
  - Research Site 1, Novara
  - Research Site 1, Parma
  - Research Site 1, Pavia
  - Research Site 1, Roma
  - Azienda Ospedaliero-Universitaria "San Giovanni Battista di Torino" Struttura Complessa Cardiologia 1, Torino
- Poland (20):
  - Research Site, Curie 1, Nysa
  - Research Site 1, Bydgoszcz, Poland
  - Research Site, Starogard Gdański, Poland
  - Research Site 1, Bydgoszcz
  - Research Site 1, Gdynia
  - Research SIte, Kielce
  - Research Site 1, Krakow
  - Research Site 2, Krakow
  - Research Site, Krakow
  - Research Site, Lubartów
  - Research Site 1, Ostrowiec Świętokrzyski
  - Samodzielny Zespol Publicznych Zakladow Opieki Zdrowotnej, Ostrołęka
  - Research Site, Pabianice
  - Samodzielnl Szpital Wojewodzki, Piotrkow Trybunalski
  - Wojewodzki Szpital Specjalistczny w Radomiu, Oddzial Kardiologil, Radom
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej, Sieradz
  - Research Site 1, Torun
  - Research Site 1, Warsaw
  - Wojskowy Instytut Medyczny, Warsaw
  - Research Site 1, Wroclaw
- Romania (5):
  - Research Site, Brasov, Romania
  - Research Site 1, Bucharest, Romania
  - Research Site 1, Tg Mures, Romania
  - Research Site 1, Bucharest
  - Research Site 1, Timișoara
- Russia (8):
  - Research Site 1, Lenskaya, Moscow
  - Research SIte 1, Moscow, Russia
  - Research Site 1, Moscow, Russia
  - Research Site, Moscow, Russia
  - Research Site 1, Saint Petersburg, Russia
  - Research Site 1, L'va Tolstogo, Sankt-Peterburg
  - Research Site 1, Solidamosty, Sankt-Peterburg
  - Research Site 1, Saint Petersburg
- Slovakia (3):
  - Research Site 1, Bratislava
  - Research Site 1, Nitra
  - Interna klinika, Fakultna nemocnica Trencin, Trenčín
- Spain (7):
  - Research Site 1, Barcelona
  - Research Site 1, Córdoba
  - Research Site 1, Madrid
  - Hospital Univeritario Virgen de la Victoria Servicio de Cardiologia, Málaga
  - Research Site 1, Málaga
  - Research Site 1, Santiago de Compostela
  - Research Site 1, Vigo
- Research Site, Geneva, Switzerland